CLINICAL TRIAL: NCT02682888
Title: Trait Anxiety Modulates Resting State Functional Connectivity of Defensive Networks
Brief Title: Trait Anxiety and Defensive Networks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, Keith Kendrick, Prof., University of Electronic Science and Technology of China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: UESTC-neuSCAN_20
Record Dates: First submitted 2016-02-08; First posted 2016-02-17 (Estimated); Last update posted 2022-02-11 (Actual); Status verified 2022-02

CONDITIONS: Healthy
Keywords: brain functional connectivity changes
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- high trait anxiety group (Experimental): experiment 1: identified according to scores of the trait anxiety scale.
  Interventions: Behavioral: trait anxiety scale
- low trait anxiety group (Experimental): experiment 1: identified according to scores of the trait anxiety scale.
  Interventions: Behavioral: trait anxiety scale
- oxytocin group (Experimental): experiment 2: intranasal administration of oxytocin
  Interventions: Drug: Oxytocin
- placebo control group (Placebo Comparator): experiment 2: intranasal administration of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Behavioral: trait anxiety scale — splitting subjects into 2 groups according to scores of the trait anxiety scale
  Arms: high trait anxiety group; low trait anxiety group
Drug: Oxytocin — intranasal administration of oxytocin
  Arms: oxytocin group
Drug: Placebo — intranasal administration of placebo
  Arms: placebo control group

SUMMARY:
to examine the association between trait and defensive network connectivity and the modulatory effect of oxytocin on it

DETAILED DESCRIPTION:
Individuals with high trait anxiety show stable anxiety proneness even in the absence of real threat, which could be a result of intrinsic hyper-connectivity in the defensive systems. In the present study, healthy subjects' trait anxiety levels will be assessed by the sub-trait inventory of the State-Trait Anxiety Inventory. Then two experiments using resting-state fMRI technique will be conducted to first map how hubs in the defensive systems organized in high anxious individuals in a stimuli-free situation (Experiment 1) and then we will examine the modulatory effect of the intranasal administration of oxytocin on functional connectivity in these independently defined defensive networks (Experiment 2).

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects without past or current psychiatric or neurological disorders

Exclusion Criteria:

* females should not be pregnant or during menstruation.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 131 (Actual)
Dates: Start 2015-12-08 (Actual); Primary Completion 2021-08-19 (Actual); Study Completion 2021-11-20 (Actual)

PRIMARY OUTCOMES:
the resting state functional connectivity changes in the defensive network | one day
  The resting-state activity can be accessed using functional magnetic resonance imaging (fMRI) by measuring spontaneous and low-frequency fluctuations (< 0.1 Hz) when the brain is at rest. Group differences will be calculated in the high trait anxiety group relative to the low trait anxiety group and in the oxytocin group relative to the placebo group.

CONTACTS AND LOCATIONS:
Overall Officials: Keith Kendrick, Dr., Principal Investigator — University of Electronic Science and Technology of China
Locations (1):
- school of life science and technology, University of Electronic Science and Technology of China, Chengdu, Sichuan, China